CLINICAL TRIAL: NCT05603455
Title: Effect of Bifidobacterium Adolescentis on Aging in Healthy Adults (45-65 Years) - a Multicenter, Double-blind, Randomized, Controlled Study
Brief Title: Effect of Bifidobacterium Adolescentis on Aging in Healthy Adults (45-65 Years)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2022-LHZHZ
Record Dates: First submitted 2022-10-19; First posted 2022-11-02 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-10

CONDITIONS: Healthy Adults (45-65 Years)

STUDY DESIGN:
Intervention Model Description: a multicenter, double-blind, randomized, controlled study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding of both the investigator (except for the investigator responsible for blinded product allocation) and the subject
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium adolescentis group (Experimental): Bifidobacterium adolescentis supplementation
  Interventions: Dietary Supplement: Bifidobacterium adolescentis
- Placebo group (Placebo Comparator): Placebo supplementation
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium adolescentis — Supplement with Bifidobacterium adolescentis twice/day in morning and tonight for 6 months
  Arms: Bifidobacterium adolescentis group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This study will include middle-aged and elderly people aged 45-65 years to carry out the translational study of Bifidobacterium adolescentis, and design a double-blind, randomized controlled clinical trial according to strict inclusion/exclusion criteria, using aging-related functional indicators, intestinal flora, DNA methylation and other advanced aging characteristic examination methods to fully and accurately assess the effects and safety of Bifidobacterium adolescentis on aging, which has the advantages of strong safety, high practice and high credibility compared with previous clinical trial protocols, laying an important foundation for improving probiotic anti-aging and exploring the development of aging intervention programs suitable for the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

1. 45-65 years of age.
2. Attending or consulting at the specialized outpatient clinics for aging diseases at 2nd Affiliated Hospital, School of Medicine, Zhejiang University and Sir Run Run Hospital, School of Medicine, Zhejiang University
3. Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

1. Known history of tumor.
2. women who are breastfeeding.
3. Those who wish to continue having children.
4. those who are unable to cooperate with investigations and testing
5. abuse of drugs, alcohol or other substances.
6. history of cardiac disease: atherosclerotic disease, heart failure, unstable angina, stable angina, etc. and chronic hypoxic diseases: emphysema, pulmonary heart disease, etc.
7. history of chronic gastrointestinal diseases (pancreatitis, IBS) and intestinal surgery.
8. endocrine disease with hyperthyroidism or cortisolism.
9. abnormal liver function, with ALT（Alanine transaminase）/AST（Aspartate aminotransferase） exceeding 2 times the upper limit of normal.
10. abnormal renal function with blood creatinine ≥ 133 μmol/L.
11. Type I diabetes or insulin-dependent type II diabetes.
12. poorly controlled chronic disease (hypertension, hyperlipidemia, type II diabetes, etc.) that is clinically unstable.
13. Vulnerable groups, including critically ill, mentally ill, cognitively impaired, minors, pregnant women, illiterate, etc.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Aging Ai 3.0 | Change from Baseline physiological age calculated by Aging Ai 3.0 at 6 months
  Calculating physiological age through physical examination indicators.The lower the physiological age calculated by Aging Ai 3.0, the better the health status.
Fasting glucose in mmol/L | Change from Baseline Fasting glucose at 6 months
  Within the normal range（3.9~6.1 mmol/L）, the health status is good
BMI（Body Mass Index）in kg/m^2 BMI | Change from Baseline BMI in kg/m^2 at 6 months
  Within the normal range, the health status is good
Epigenetic clock | Change from Baseline physiological age calculated by Epigenetic clock at 6 months
  physiological age was calculated by Epigenetic clock through DNA methylation.The lower the physiological age calculated by Epigenetic clock, the better the health status.
Bone density in g/cm^3 | Change from Baseline Bone density in g/cm3 at 6 months
  The higher the Bone density, the better the health status
Triglycerides in mmol/L | Change from Baseline Triglycerides at 6 months
  Within the normal range（2.26~5.6 mmol/L）, the health status is good
Cholesterol in mmol/L | Change from Baseline Cholesterol at 6 months
  Within the normal range（3.6~5.2 mmol/L）, the health status is good
Telomere level | Change from Baseline Telomere level at 6 months
  Telomere level was detected by qRT（quantitative real-time）-PCR（Polymerase Chain reaction）. The lower the Cycle Threshold，the higher the Telomere level，which means the healthier and younger.
Blood pressure | Change from Baseline Systolic Blood Pressure and diastolic blood pressure at 6 months
  Within the normal range, the health status is good
body fat percentage | Change from Baseline body fat percentage at 6 months
  The higher the body fat percentage, the better the health status
Markers for cell senescence | Change from Baseline the expression level of indicators at 6 months
  The expression level of Markers for cell senescence was detected by qRT（quantitative real-time）-PCR（Polymerase Chain Reaction）.The higher the Cycle Threshold，the lower the expression level of Markers for cell senescence, which means the healthier.

SECONDARY OUTCOMES:
Flora Clock | Change from Baseline physiological age calculated by Flora Clock at 6 months
  Calculating physiological age through intestinal flora.The lower the physiological age calculated by Flora Clock, the better the health status.
Mini-Nutritional Assessment | Change from Baseline score at 6 months
  The score (0-30)was calculated by Mini-Nutritional Assessment. The higher score calculated by Mini-Nutritional Assessment means a better outcome
The Medical Outcomes Study Short Form 36(SF-36) | Change from Baseline score at 6 months
  The score (36-145)was calculated by The Medical Outcomes Study Short Form 36. The higher score calculated by The Medical Outcomes Study Short Form 36 means a better outcome
Pittsburgh sleep quality index | Change from Baseline score at 6 months
  The score (0-21)was calculated by Pittsburgh sleep quality index The higher score calculated by Pittsburgh sleep quality index means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: liangjing wang, doctor, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Sir RUN RUN Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided